CLINICAL TRIAL: NCT05139745
Title: Histological Evaluation of BTL-899 Device´s Effect on Fat Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BTL-899_CTUS400
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Fat Burn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Histological evaluation of BTL-899 device´s effect on fat tissue (Experimental): This group will be treated with 100% of the treatment parameter settings
  Interventions: Device: BTL-899
- Sham treatment (Sham Comparator): This group will be treated with 5% of the treatment parameter settings
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — BTL-899 treatment

SUMMARY:
This study will evaluate the safety and performance of the BTL-899 device for non-invasive treatment of subcutaneous fat. The changes in the fat tissue related to the activity of caspase-3 will be assessed histologically. The study is a prospective single-center single-blinded two-arm study. The subjects will be enrolled and assigned into two study groups; Group A which will receive active treatment and Group B which receives sham treatment and will serve as a control to verify the treatment outcomes. Subjects will be required to complete only one (1) treatment visit and three (3) follow-up visits (at 8 hours, 24 hours and 7 days post treatment). All of the study subjects will receive the treatment (either active or sham) with the subject device.

At the baseline visit, health status will be assessed. Inclusion and exclusion criteria will be verified and informed consent will be signed. Punch biopsies from the treated abdominal area will be taken to examine the changes related to caspase-3 activity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study.
* Willingness to abstain from partaking in any treatments other than the study procedure
* Willingness to comply with study instructions, to return to the clinic for the required visits and to undergo punch biopsies in the abdominal area.

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants in the treated area
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles in the treated area
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations in the treated area
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Application during pregnancy, postpartum period, nursing, and menstruation
* Graves' disease
* Skin related autoimmune diseases that may contradict the biopsy
* Poor healing and unhealed wounds in the treatment area
* Any disease or condition contradicting the skin tissue biopsy
* Any disease or condition that may compromise the histologic observation at the pathologist discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Increased caspase-3 activity | 1 month
  Biopsy samples of the abdominal fat tissue will be processed for histological evaluation by a certified laboratory. Conventional staining will be used to determine the changes in the fat tissue related to the increase in caspase-3 activity, which is associated with elevated levels of fat tissue apoptosis, and to examine other morphological changes of treated tissue, in all collected samples. Post-treatment findings will be compared to the baseline. The results of both study groups will be compared as well.

SECONDARY OUTCOMES:
Safety assessment | 1 month
  Occurrence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Laser and Surgery Specialist, a Division of Schweiger Dermatology, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No